CLINICAL TRIAL: NCT02075502
Title: A Community-based Exercise Program to Improve Walking Outcomes in Patients With Peripheral Artery Disease
Brief Title: Community Walking Exercise for Patients With Peripheral Artery Disease
Acronym: GAIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mays-1; 1K01HL115534 (NIH)
Record Dates: First submitted 2014-02-13; First posted 2014-03-03 (Estimated); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Peripheral Artery Disease
Keywords: claudication; community walking exercise; community-based participatory research; exercise adherence; endovascular therapy
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Exercise therapy (Experimental): Claudication, no peripheral revasc
  Interventions: Behavioral: Exercise therapy
- Exercise advice (Placebo Comparator): Claudication, no peripheral revasc
  Interventions: Behavioral: Exercise therapy
- lower extremity ET, exercise therapy (Experimental)
  Interventions: Behavioral: Exercise therapy; Procedure: lower extremity ET
- lower extremity ET, exercise advice (Placebo Comparator)
  Interventions: Procedure: lower extremity ET
- Peripheral open intervention, exercise therapy (Experimental)
  Interventions: Behavioral: Exercise therapy; Procedure: peripheral open intervention
- Peripheral open intervention, exercise advice (Placebo Comparator)
  Interventions: Procedure: peripheral open intervention

INTERVENTIONS:
Behavioral: Exercise therapy — The exercise therapy program with training, monitoring and coaching enhanced by community-based participatory research (CBPR) (TMC+) is a comprehensive approach to community-based walking exercise for improving PAD patient outcomes. The components of TMC+ are optimal training guidelines for patients (i.e., T), monitoring from both investigators and patient self-monitoring (i.e., M), coaching from investigators on how to improve patients' walking ability (i.e., C), and finally enhancements from CBPR practices (+).
  Arms: Exercise advice; Exercise therapy; Peripheral open intervention, exercise therapy; lower extremity ET, exercise therapy
Procedure: lower extremity ET — catheter-based revascularization of peripheral arteries (background treatment part of standard clinical care at hospital)
  Arms: lower extremity ET, exercise advice; lower extremity ET, exercise therapy
Procedure: peripheral open intervention — revascularization of lower extremities with open bypass surgery (background treatment part of standard clinical care at hospital)
  Arms: Peripheral open intervention, exercise advice; Peripheral open intervention, exercise therapy

SUMMARY:
The primary aim of the study is to determine the effect of a community-based walking exercise program with detailed training, monitoring, and coaching (TMC) exercise components enhanced by community-based participatory research (CBPR) practices (TMC+) on the primary outcome of peak walking time (PWT) in patients with peripheral artery disease (PAD).

DETAILED DESCRIPTION:
The investigators will test the hypothesis that PAD patients randomized to the exercise program in the community setting incorporating TMC+ will improve walking ability compared with patients who receive the standard of care (exercise advice). Secondary hypotheses include a significant improvement in patient-reported outcomes, an improvement in functional ability or a significant increase in volume of physical activity for patients who complete community-based walking exercise when compared with patients receiving the standard of care. Exploratory hypotheses include a significant improvement in PWT for 1) patients receiving a combination of lower extremity endovascular therapy (ET) and community-based walking exercise or 2) open peripheral intervention and community-based walking exercise compared to patients who do not receive endovascular therapy or open intervention and receive only the standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with atherosclerotic PAD
* ≥40 years of age
* An abnormal ankle-brachial index (ABI) of ≤.90
* For patients with an ABI >.90 and <1.00, a post-exercise ABI drop of 15% or more compared to the resting ABI
* Patients receiving lower extremity ET or peripheral open intervention
* Patients not receiving lower extremity ET or peripheral open intervention but present with stable claudication and an abnormal ABI

Exclusion Criteria:

* Lower extremity amputation(s), including a toe amputation, which interfere (s) with walking on the treadmill
* Individuals with critical limb ischemia defined by ischemic rest pain or ischemic ulcers/gangrene on the lower extremities
* PAD of non-atherosclerotic nature (e.g., fibromuscular dysplasia, irradiation, endofibrosis)
* Coronary artery bypass grafts or major surgical procedures within 6 months prior to screening
* Individuals whose walking exercise is primarily limited by symptoms of chronic obstructive pulmonary disease, angina, or heart failure
* Individuals who are unable to walk on the treadmill at a speed of at least 2 mph for at least 1 minute
* Individuals who have had a myocardial infarction within 3 months prior to screening
* Individuals who demonstrate symptoms consistent with acute coronary syndrome
* Individuals who exhibit ischemia as documented on the 12-lead electrocardiogram including horizontal or down-sloping ST-segment depression ≥0.5 mm at rest and >1 mm with exercise in 2 contiguous leads, relative to the PR-segment (ST-segment measured 0.08 seconds after the J point, ST-segment elevation ≥1 mm)
* Individuals who have had a transient ischemic attack or stroke 3 months prior to screening
* Individuals with left bundle branch block or sustained ventricular tachycardia (>30 sec) during screening
* Individuals with uncontrolled hypertension (≥180 systolic or ≥100 diastolic resting blood pressure) during screening
* Treatment with pentoxifylline or cilostazol for the treatment of claudication 4 weeks prior to screening; Patients can be reconsidered for study inclusion following a 1 month washout period from these medications
* Electrolyte abnormalities (e.g., potassium <3.3 mmol∙Lˉ1 )
* Pregnancy, fertility without protection against pregnancy (for women of childbearing potential, a serum pregnancy test will be performed at screening)
* Incarcerated individuals
* Individuals acutely impaired by alcohol or other illicit drugs
* Poorly controlled diabetes defined as glycated hemoglobin >12%
* Severely anemic patients (Hgb <11 g∙dLˉ1 for women and <10 g∙dLˉ1 for men)
* For patients who have not received peripheral revascularization, an ABI of >0.90
* For patients with equivocal resting ABIs (0.91-0.99), a drop of <15% in the post-exercise ABI
* For individuals with non-compressible vessels (ABI >1.39) who have a toe- brachial index (TBI) >0.70
* Inability to speak English
* Other clinically significant disease that is, in the opinion of the study team, not stabilized or may otherwise confound the results of the study

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2014-02-01 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Change in peak walking time (PWT) | Baseline, post-revascularization (ET or open intervention) (4 weeks, if applicable), post-12 weeks (exercise and control groups), 6 months following intervention time period

SECONDARY OUTCOMES:
Change in claudication onset time (COT) | Baseline, post-revascularization (ET or open intervention), post-12 weeks (exercise and control groups), 6 months following intervention time period
Change in patient-reported outcomes | Baseline, post-revascularization (ET or open intervention), post-12 weeks (exercise and control groups), 6 months following intervention time period
Change in peak oxygen uptake | Baseline, post-revascularization (ET or open intervention), post-12 weeks (exercise and control groups), 6 months following intervention time period
Change in functional ability | Baseline, post-revascularization (ET or open intervention), post-12 weeks (exercise and control groups), 6 months following intervention time period
  Functional ability will be assessed with the 6-min walk test and Short Physical Performance Battery which consists of 1) walking short distances, 2) completing balance tests and 3) sit and standing from a chair 5 times.
Evaluation of total volume of activity | post-12 weeks (exercise and control groups)
Evaluation of exercise adherence | post-12 weeks (exercise and control groups)
  For patients randomized to the exercise therapy group

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J. Mays, PhD, MPH, MS, Principal Investigator — International Heart Institute of Montana Foundation
Locations (1):
- International Heart Institute of Montana Foundation, Missoula, Montana, United States

REFERENCES:
- See also: Click here for more information about the sponsor. — http://www.nhlbi.nih.gov/
- See also: Click here for more information about the sponsor. — http://www.nih.gov/

DOCUMENTS (1):
  • Informed Consent Form (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/02/NCT02075502/ICF_000.pdf